CLINICAL TRIAL: NCT05415436
Title: Analyzing the Relationship Between Rate of Induction and Perioperative Hypotension Using Propofol
Brief Title: Analyzing the Relationship Between Speed Propofol is Given and Low Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Propofol study
Record Dates: First submitted 2022-04-20; First posted 2022-06-13 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-12

CONDITIONS: Hypotension on Induction

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A- propofol given at FDA approved administration speed (No Intervention)
- Group B- propofol given over 120 seconds (Experimental)
  Interventions: Other: Propofol slow administration

INTERVENTIONS:
Other: Propofol slow administration — Propofol will be slowly administered over 120 seconds by anesthesia provider
  Arms: Group B- propofol given over 120 seconds

SUMMARY:
The objective of this study is to evaluate the hemodynamic changes related to Propofol administration rate. We hypothesize that slow administration of IV propofol will have less hemodynamic disturbances and will require less amount of vasoactive medication for BP correction when compared to standard FDA approved administration rate.

ELIGIBILITY:
Inclusion Criteria:

* any patient from 18 till 80 years of age
* patient undergoing non-cardiac elective surgery
* duration of the surgery longer than one hour
* native/fluent English speaker
* patients whose staff anesthesiologist planned to use Propofol as a primary anesthetic for induction

Exclusion Criteria:

* any patient admitted for non-elective surgery
* any patient undergoing cardiac surgery
* any patient under 18 years of age
* any patient older than 80 years of age
* any patient with history of severe heart disease (CHF with significant limitations of activity due to sever symptoms, prior heart surgery, atrial fibrillation, etc.)
* any patient with pre-operative hemodynamic instability (e.g. sepsis, chronic kidney disease, liver cirrhosis) who requires constant or intermittent administration of vasoactive or inotropic medication to support vital signs (BP)
* any patient on vasoactive or inotrop medications in early pre-operative period (within 24 hours prior to the surgery)
* any patient who does not speak English or not fluently
* any patient with cognitive impairment or mentally incapacitation
* any pregnant or breastfeeding females
* any patient whose staff anesthesiologist planned to use a primary anesthetic other than Propofol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Pappada, PhD, Principal Investigator — University of Toledo
Locations (1):
- The University of Toledo Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A- Propofol Given at FDA Approved Administration Speed: propofol given at FDA approved administration speed
Period: Overall Study
Arm/Group | Group A- Propofol Given at FDA Approved Administration Speed | Group B- Propofol Given Over 120 Seconds
Started | 54 | 46
Completed | 52 | 46
Not Completed | 2 | 0
Not completed — Surgeon cancelled procedure | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A- Propofol Given at FDA Approved Administration Speed | Group B- Propofol Given Over 120 Seconds | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 32 | 68
  >=65 years | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 24 | 21 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 54 | 46 | 100

OUTCOME MEASURES:

1. Primary Outcome: Patients Administered Propofol at a Slower Rate of Infusion Will Have Lower Incidence of Post Induction Hypotension Than Patients Administered Propofol at FDA Approved Rate.
Description: We will collect the patient's blood pressure intra-operatively every 5 minutes starting on induction up to one hour after induction and compare.
Time Frame: induction to 1 hour post induction
Measure: Count of Participants; unit: Participants
Arm/Group | Group A- Propofol Given at FDA Approved Administration Speed | Group B- Propofol Given Over 120 Seconds
Number analyzed (Participants) | 53 | 46
Participants
  Number of participants with post induction hypotension | 4 | 2
  Number of participants without post induction hypotension | 49 | 44

2. Secondary Outcome: Patients Administered Propofol at a Slower Rate Will Have Less Complications During the Early Post-op Period Than Patients Administered Propofol at FDA Approved Rate.
Description: We will collect the patient's blood pressure post-operatively and length of hospital stay and compare.
Time Frame: immediate post-op to 30 days post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group A- Propofol Given at FDA Approved Administration Speed | Group B- Propofol Given Over 120 Seconds
Number analyzed (Participants) | 53 | 46
Participants
  Participants requiring albumin administration | 4 | 0
  Participants requiring vasopressin administration | 4 | 0

ADVERSE EVENTS:
Time Frame: Data was collected from date of enrollment in the study, which was the patient's procedure date, to 30 days post-operatively.
Arm/Group | Group A- Propofol Given at FDA Approved Administration Speed | Group B- Propofol Given Over 120 Seconds
All-Cause Mortality (participants affected / at risk) | 1/53 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/53 | 0/46
Other Adverse Events (participants affected / at risk) | 0/53 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A- Propofol Given at FDA Approved Administration Speed (N=53) | Group B- Propofol Given Over 120 Seconds (N=46)
participant died 5 days post study procedure due to multi system organ failure (Vascular disorders) | 1 (1) | 0 (0) — investigator determined that cause of death was unrelated to study procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT05415436/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT05415436/ICF_001.pdf